CLINICAL TRIAL: NCT01788865
Title: Efficacy and Safety of a Covered Self-expandable Dual-layered Metallic Mesh Stent (UVENTA™) in Ureteral Obstruction: Prospective, Multi-center, Open Label Study
Brief Title: Efficacy and Safety of a Covered Self-expandable Dual-layered Metallic Mesh Stent (UVENTA) in Ureteral Obstruction
Acronym: UVENTA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, HAN, DEOK HYUN, HAN, DEOK HYUN, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URT-001
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Ureteral Obstruction
Keywords: covered Metal stent; ureteral obstruction
MeSH Terms: conditions — Ureteral Obstruction | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cSEMS (Experimental): Patients with malignant ureteral obstruction have cSEMS(Covered self-expandable dual-layered metal stent) implant
  Interventions: Device: cSEMS(Covered self-expandable dual-layered metal stent) implant

INTERVENTIONS:
Device: cSEMS(Covered self-expandable dual-layered metal stent) implant
  Other Names: UVENTA™ Ureteral Stent, Taewoong medical

SUMMARY:
The purpose of this study is to evaluate Efficacy and Safety of a covered self-expandable dual-layered metallic mesh stent (UVENTA) in ureteral obstruction.

DETAILED DESCRIPTION:
Prospective, Multi-center, open label, single arm Study

1. Treatment

   - Covered self-expandable dual-layered metallic mesh Stents(cSEMS) are implanted in patents with malignant ureteral obstruction
2. Follow up

   * Assessments including X-ray(KUB), are done 3, 6, 12, 18 and 24 months after the procedure.
   * Diuretic RI scan (DTPA, MAG-3) 3, 6, 12 months after the procedure
   * Imaging such as IVP(Intravenous Pyelogram), ultrasonogram, CT(Computed Tomogram) are performed at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily agree to participation and submitted a written informed consent for this study, and 20~80 years
2. One out of following cases below apply to Patients who have malignant ureteral obstruction or have benign ureteral obstruction without improvement after previous treatment

   * Patients who doesn't want to have regular replacement of plastic stent
   * Patients who has no improvement of obstruction after plastic stent implant
   * Patients who want other Urinary diversion because of stimulatory sign or pain due to plastic stent
3. Patients with no previous ureteral metal stenting procedure experience.
4. Patients with more than 6 months of life expectancy
5. Patients understanding the objective of the study and who are willing to sign a consent

Exclusion Criteria:

1. Patients with Urothelial Carcinoma
2. Patients with bladder invasion of malignant tumor
3. Patients with bladder dysfunction or obstruction of lower urinary tract
4. one or more times Recurrent Urinary stone in the last 3 years
5. 2 or more times upper urinary tract infection without upper urinary tract obstruction
6. Karnofsky scores < 60
7. Patients with Bacteriuria
8. Inadequate Patient to participate in the study as judged by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months
  Rate of Ureter units maintaining patency without interventions after technical success of the primary procedure(Diuretic RI scan: T½ < 20 min)

SECONDARY OUTCOMES:
Technical success rate | 1week, 1 month
  Rate of technical success(each Ureter) resolving the stenosis and passing the contrast medium from the kidney to urinary bladder
Final patency rate | 12 months
  Rate of Ureter units maintaining patency without interventions aside from re-stenting(investigational device) after technical success of the primary procedure(Diuretic RI scan: T½ < 20 min)
Adverse Event | 1week, 1, 3, 6, 9, 12 months
  Rate of total Adverse Events and Adverse Events relevant to Investigational Device
Predictive Risk Factors for Primary patency rate | 12 months
  Age, Sex, type of tumor(benign/malignant), length of stenosis, location of stenosis, UVJ cross, balloon catheterization, etc.
the primary patency rate among different location of distal stent | 12 months
  difference of the primary patency between the group of Distal stent located in urinary bladder and ureter
Ureteral stent symptom questionnaire(USSQ) | 1, 3, 6, 9, 12 months
  Comparative analysis of USSQ : before procedure and after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Deok Hyun Han, M.D., Principal Investigator — Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine; Hyeong keun Park, M.D. Ph.D., Principal Investigator — Department of Urology, Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul